CLINICAL TRIAL: NCT03506126
Title: Determination of Leucine Requirement in Adults Over 60 Years of Age Using the Indicator Amino Acid Oxidation Method
Brief Title: Requirement for Leucine in Adults Over 60 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Principal Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000059679
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: amino acid requirement; elderly; leucine; dietary requirement
MeSH Terms: interventions — Leucine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Leucine Adults > 60 (Experimental): In this arm, all subjects will receive all 8 of the leucine test levels, assigned in random order.
  Interventions: Other: Leucine

INTERVENTIONS:
Other: Leucine — There are 8 different leucine test levels ranging from 20 to 120 mg of leucine per kilogram body weight per day (20-120 mg/kg/d)

SUMMARY:
This study aims to determine the requirement for leucine, an essential amino acid, in adults over the age of 60 years. It is known that protein and amino acid metabolism may be altered with age and leucine, in particular, may be important in the diet of older adults.

Eight different levels of leucine intake will be tested in each subject in random order. Each level of leucine intake will involve a 3-day maintenance diet, with measures being collected on the third.

DETAILED DESCRIPTION:
Leucine is an essential amino acid that is an important component of protein and stimulator of muscle protein synthesis. It is known that as people get older, over the age of 60, our body goes through many changes such as increase in fat mass and decrease in lean mass such as muscle. This is why we are studying how much of the essential amino acid, leucine, the body needs at this particular age.

The indicator amino acid oxidation (IAAO) method is a minimally invasive method for determining essential amino acid requirements.

As essential amino acids cannot be stored in the body, they are either partitioned into protein synthesis or oxidized if in excess. The premise of the IAAO is that when any essential amino acid is limiting in the body then all other amino acids lose their ability to contribute to protein synthesis and are instead oxidized. The method therefore involves providing graded intakes (from deficient to excess) of the test amino acid, leucine, and then measuring the oxidation of another amino acid, which is called the indicator amino acid. This is done by isotopically labelling the indicator amino acid (we often use 13C- phenylalanine) and then measuring the appearance of labelled carbon dioxide (13CO2) in breath with the different intakes of the test amino acid, leucine. The requirement for leucine will be determined by the "breakpoint" - the point at which oxidation of 13C- phenylalanine will plateau.

For the study, subjects will first participate in a pre-study assessment in which height, weight, body composition (fat mass and muscle mass) and resting energy expenditure and medical history will be assessed. Also, 10 ml of blood will be collected to test for diabetes and kidney function. The purpose of the pre-assessment is to calculate subject's dietary requirements for the study, and to assess health status, activity level and dietary patterns.

Subjects will then participate in up to 8 different 3-day studies that will be separated by a minimum of 1 week between each 3-day study. The first 2 days are adaptation days and subjects will consumed the maintenance diet at home s 4 equal meals. The 3rd day is called a study day and subjects will consumed 8 hourly formulas; the first 3 at consumed at home and the remaining 5 are consumed at the Clinical Research Centre at the Hospital for Sick Children. Immediately after the 4th meal, 4 baseline breath and 3 baseline urine samples are collected. After the 5th meal, rate of carbon dioxide production (VCO2) is measured by indirect calorimetry for a period of 20 minutes. The 5th, 6th, 7th, and 8th meal will contain a small amount of isotope labelled phenylalanine (13C phenylalanine). Two and a half hours after the isotope (13C phenylalanine) is given, 4 plateau breath and 3 plateau urine samples are collected.

Breath samples are used to measure the enrichment of isotopic labelled CO2 (13CO2). Urine samples are used to measure the enrichment of isotopic labelled phenylalanine (13C phenylalanine). Through a series of calculations and applying a two-phase regression analysis, we will be able to determine the requirement for leucine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males > 60 years
* Willingness to participate in the study and completed the screening procedures (height, weight, fasting blood sample and medical history questionnaire).
* No recent history of weight loss
* Absence of chronic disease or acute illness that could affect protein and AA metabolism (diabetes, cancer, liver or kidney disease, HIV, acute cold or flu, hypo or hyperthyroidism, rheumatoid arthritis treated with anti-inflammatory medications).
* Non-smoking
* Willingness to consume the diet provided

Exclusion Criteria:

* Presence of disease known to affect protein and AA metabolism (diabetes, cancer, liver or kidney disease, HIV, acute cold or flu, hypo or hyperthyroidism, rheumatoid arthritis treated with anti-inflammatory medications).
* On medications known to affect protein and amino acid metabolism (steroids).
* Recent significant weight loss.
* Individual on weight reducing diets.
* Inability to tolerate the diet
* Unwilling to have blood drawn from a venous access, or using a ventilated hood indirect calorimeter for the purposes of the study.
* Significant coffee consumption of more than 2 cups/day
* Significant alcohol consumption of more than one drink/day

Min Age: 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Determination of leucine requirement in adults over 60 y | 3 years
  Rate of 13C-phenylalanine oxidation.

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szwiega S, Pencharz PB, Rafii M, Lebarron M, Chang J, Ball RO, Kong D, Xu L, Elango R, Courtney-Martin G. Dietary leucine requirement of older men and women is higher than current recommendations. Am J Clin Nutr. 2021 Feb 2;113(2):410-419. doi: 10.1093/ajcn/nqaa323. PMID 33330915